CLINICAL TRIAL: NCT03362619
Title: Innovative Treatment of Cervical Cancer Using Engineered Antigen-specific Immune Effectors (EIEs)
Brief Title: Engineered Immune Effectors Against Cervical Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Principal Investigator, Lung-Ji Chang, President, Shenzhen Geno-Immune Medical Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-17019
Record Dates: First submitted 2017-11-20; First posted 2017-12-05 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Cervical Cancer
Keywords: Cervical cancer; Cytotoxic lymphocyte; CC-CTL
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CC-EIEs (Experimental): Autologous cervical cancer specific engineered immune effectors (EIEs)
  Interventions: Biological: CC-EIEs

INTERVENTIONS:
Biological: CC-EIEs — 2 to 4 infusions, once a week, for 1x10^5~1x10^7 CTLs/kg via IV, abdominal cavity or intratumoral injection each time

SUMMARY:
The primary objective of this study is to evaluate the safety of cervical cancer specific engineered immune effectors (CC-EIEs). The secondary objectives are to evaluate the rate of successful CC-EIE generation in vitro and determine the anti-CC efficacy.

DETAILED DESCRIPTION:
Cervical cancer (CC) is a cancer arising from the cervix. Human papillomavirus (HPV) infection causes more than 90% of the cases. Other risk factors include smoking, a weak immune system, birth control pills, starting sex at a young age, and having many sexual partners, but these are less important. Worldwide, CC is both the fourth-most common cause of cancer and the fourth-most common cause of death from cancer in women. The treatment of CC consists of surgical intervention, radiation, chemotherapy and immunotherapy.

Adoptive immunotherapy with cytotoxic T lymphocytes reactive with specific viral antigens has proven to be effective. Here, the investigators aim to evaluate the safety and efficacy of multiple infusions of CC-specific engineered immune effectors including cytotoxic T lymphocytes in patients.

ELIGIBILITY:
Inclusion Criteria:

1. Written, informed consent obtained prior to any study-specific procedures.
2. Age older than 10 years.
3. Eastern Cooperative Oncology Group (ECOG) PS of 0 or 1.
4. Expected survival ≥ 12 weeks.
5. Not pregnant, and on appropriate birth control if of childbearing potential.
6. Evidence of high-risk HPV infection.
7. Stage III-IV or recurrent cervical cancer.
8. Initial hematopoietic reconstitution with

   * neutrophils (ANC) ≥ 1,000/mm^3;
   * platelet (PLT) ≥ 100,000/mm^3.
9. Proper renal and hepatic functions (ULN denotes "upper limit of normal range") with

   * serum creatinine ≤ 2×ULN;
   * serum bilirubin ≤ 2×ULN;
   * AST/ALT ≤ 2×ULN;
   * ALKP ≤ 5×ULN;
   * serum bilirubin. 2.0 is acceptable in the setting of known Gilbert's syndrome.
10. Human immunodeficiency virus (HIV) and Hepatitis C virus (HCV) test negative.

Exclusion Criteria:

1. Patients with

   * cervical benign lesions: cervical columnar epithelium ectopic, cervical polyps, cervical endometriosis and cervical tuberculous ulcers;
   * cervical benign tumors: cervical submucous myoma, cervical cancer, cervical papilloma.
2. Patients with evidence of abdominal free air not explained by paracentesis or recent surgical procedure (prior, current or planned treatment).
3. Previous exposure to mouse SCC antibody.
4. Current or recent treatment (within the 28-day period prior to Day 0) with another investigational drug or previous participation in this study.
5. Minor surgical procedures within 2 days prior to Day 0 (including central venous access device placement for chemotherapy administration, tumor biopsies, needle aspirations).
6. Pregnant or lactating females.
7. Inadequate bone marrow function with

   * absolute neutrophil count < 1,000/mm^3;
   * platelet count < 100,000/mm^3;
   * Hb < 9 g/dL.
8. Inadequate liver and renal function with

   * serum (total) bilirubin > 1.5 x ULN;
   * AST & ALT > 2.5 x ULN (> 5 x ULN in patients with liver metastases);
   * alkaline phosphatase > 2.5 x ULN;
   * serum creatinine >2.0 mg/dl (> 177 μmol/L);
   * urine dipstick for protein uria should be < 2+. Patients with ≥ 2+ proteinuria on dipstick urinalysis at baseline should undergo 24 hour urine collection and must demonstrate < 1 g of protein/24 hr.
9. Serious active infection requiring i.v. antibiotics at during screening.
10. Subject actively infected with HCV (HCV antibody positive), HBV (HBsAg positive), HIV (HIV antibody positive), HTLV (HTLV antibody positive), Treponema pallidum antibody positive or TB culture positive.

Ages: 10 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-11-15 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Safety of CC-EIEs in patients using CTCAE version 4.0 standard to evaluate the level of adverse events | 6 months
  Physiological parameter (measuring cytokine response, fever, symptoms)

SECONDARY OUTCOMES:
Functional analyses of CC-EIEs in vitro | 4 weeks
  The specificity of CC-EIEs in vitro will be analysed by enzyme-linked immunospot assay (ELISPOT).
Anti-tumor effects | 1 year
  Objective response, such as complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD) will be assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Lung-Ji Chang, PhD, Principal Investigator — Shenzhen Geno-Immune Medical Institute; Qichun Cai, MD, Study Director — Jinshazhou Hospital of Guangzhou University of Chinese Medicine; Xun Lai, MD, Study Director — Yunnan Cancer Hospital & The Third Affiliated Hospital of Kunming Medical University & Yunnan Cancer Center
Locations (3):
- China (3):
  - Jinshazhou Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong
  - Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong
  - Yunnan Cancer Hospital & The Third Affiliated Hospital of Kunming Medical University & Yunnan Cancer Center, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: No